CLINICAL TRIAL: NCT01810328
Title: Validation of a Genomics Based Prognostic in Severe Trauma
Brief Title: A Validation of a Genomics Based Prognostic in Severe Trauma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of General Medical Sciences (NIGMS) (NIH); Massachusetts General Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB201601501-N; R01GM104481-01 (NIH); 482-2012 (Other: University of Florida)
Record Dates: First submitted 2013-03-11; First posted 2013-03-13 (Estimated); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Trauma; Complications; Multiple Organ Failure
MeSH Terms: conditions — Wounds and Injuries; Multiple Organ Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traumatized population (Active Comparator): In the traumatized population (severe blunt traumatic injury), blood samples will be collected at admission, days 1, 4, 7, 14, 21 and 28, or until discharge from the ICU or death. A total of 5 mLs of blood will be collected at admission and day 1, 4 mLs of blood will be collected at each remaining time point.
  Interventions: Other: Traumatized population
- Healthy Volunteers (Active Comparator): The healthy volunteer participants will donate a one-time 5 mL blood sample which will undergo rapid leukocyte genomic screening. These controls will allow the investigators to determine if the values obtained are accurate, reliable, and repeatable.
  Interventions: Other: Healthy Volunteers

INTERVENTIONS:
Other: Traumatized population — In the traumatized population (severe blunt traumatic injury), blood samples will be collected at admission, days 1, 4, 7, 14, 21 and 28, or until discharge from the ICU or death. A total of 5 mLs of blood will be collected at admission and day 1, 4 mLs of blood will be collected at each remaining time point.
  Arms: Traumatized population
Other: Healthy Volunteers — The healthy volunteer participants will donate a one-time 5 mL blood sample which will undergo rapid leukocyte genomic screening. These controls will allow the investigators to determine if the values obtained are accurate, reliable, and repeatable.
  Arms: Healthy Volunteers

SUMMARY:
The purpose of this study is to learn more about how to treat patients with severe injuries related to trauma and to prevent failure of vital organs in this patient population. Approximately 200 severely injured patients with blunt trauma and 40 healthy volunteer subjects will be enrolled in this study. During the study seven blood samples (4-5 mls) will be collected from patients who have suffered severe trauma over a 28 day period. A one time 5 ml blood sample will be collected from the healthy volunteers. Clinical data will be collected daily while patients are hospitalized. The initial blood sample must be collected from qualifying patients within the first 12 hours of admission to the hospital. The reason for blood sampling is to validate a rapid genomic test in real time. Once confirmed, this genomic test can be used to identify patients who will have a complicated clinical course and would, therefore, be good candidates for interventional, immunomodulatory therapies.

DETAILED DESCRIPTION:
Specific Aim: To prospectively validate a rapid genomic test obtained from blood leukocyte subpopulation of severely traumatized patients in the first 24 hours after admission, that can be used to discriminate those patients who will have a complicated clinical trajectory and would, therefore, be good candidates for interventional, immunomodulatory therapies.

Following severe blunt traumatic injury and during recovery, alterations in the leukocyte transcriptome occur. Thus, we propose that a leukocyte transcriptome signal based on the expression of the validated 63 total leukocyte or 181 PMN genes can be used to identify patients who are at risk of a complicated clinical outcome, either alone or when combined with anatomical or physiological predictors. The goal of this clinical trial is to validate the predictive ability of this transcriptome-based prognostic.

This is a non-interventional, observational study of 200 severely injured patients with blunt trauma and 40 healthy volunteers. The entry criteria will be the same as has been used for the past eight years with the Glue Grant. Severe blunt injured patients that meet the inclusion criteria will undergo rapid leukocyte genomic screening at admission and the following morning(~24 hrs). Additional blood samples will be collected at 4, 7, 14, 21 and 28 days, or as long as the patients are in the trauma or surgical intensive care unit, for banking.

Over a four year period, we will enter 240 subjects from the University of Florida and from the University of Washington at Harborview Medical Center. In the trauma subjects, blood samples will be collected at admission, days 1, 4, 7, 14, 21 and 28, or until discharge from the ICU or death. A total of 4 to 5 mLs of blood will be collected at each time point. In the healthy volunteers, a one-time blood sample will be collected.

Screening and Consent: Trauma patients will be identified by study personnel following presentation to the emergency room. The subject or legal next-of-kin will be approached for consent within 96 hours if the patient meets entry criteria. We ask for delayed consent in this patient population for 96 hours due to the severity of the injuries, the vulnerable nature of the patient at this early time, and the challenge in reaching the patient's legal representatives. Should informed consent not be obtained within 96 hours, all blood samples and data collected will be discarded.

Healthy volunteer subjects will be identified from the general population by way of advertisement flyers posted at the respective universities. The flyers will provide contact information for the laboratories. Healthy subjects will be screened via inclusion/exclusion criteria upon contact. If appropriate for participation, the subject will be consulted for consent.

Blood will be collected from existing access, or by venipuncture, if required. Blood will be promptly placed on ice and transferred to the laboratory where it will be processed for cell lysates and plasma.

All other relevant clinical data and hemodynamic measurements will be collected daily while patient is hospitalized.

* Demographic information.
* Past and present medical records
* Laboratory, microbiology, and all other test results
* X-ray, CT, MRI, US and all other imaging test results
* Records about any medication received during admission
* Records of physical exam during admission
* Records of all vital signs and hemodynamic monitoring during admission
* Records of any procedure or intervention during admission
* Records of any procedure or intervention during hospital admission
* Condition at the discharge and discharge facility

Each of the two clinical sites will maintain responsibility for the collection and storage of clinical data. REDCap (Research Electronic Data Capture) will be used for the collection of clinical data. It is a secure, Web-based application designed to support traditional case report form data capture. Cell lysates obtained at the University of Washington-Harborview Medical Center will be shipped to the University of Florida for genomic analyses, while plasma samples collected at Shands Hospital at the University of Florida will be shipped to the University of Washington for cytokine analyses by Luminex™. At yearly intervals, electronic data transfers from the University of Florida to the University of Washington of both non-identifiable, coded clinical data and cytokine and genomic data will occur.

Blood draws related to the study will be done at the bedside in a manner compatible with the standard of clinical care or in our laboratories for healthy volunteers. Tubes used for the blood draws related to study will be labeled with the unique study number and will not carry any patient identifier. The key linking unique patient number and patients personal identifiers will be stored in a password protected and encrypted file and will be only accessible for the PI and the research team. All patient collected clinical data will be stored in a cabinet that is located in the office of the PI or research team. The computer used for the storage of data will be located in the office of the PI or research staff that is always locked. The computer will be password protected and encrypted.

We have based our assessment for the number of subjects on our preliminary data set from 1637 severe trauma subjects. In that study, of the 1637 subjects, 31% or 507 patients had a time to recovery of less than five days, and could be identified as having an uncomplicated outcome. In contrast, 442 patients or 27% had complicated outcome, as defined by either late death or MOF lasting longer than 14 days. Assuming a similar frequency of complicated and uncomplicated patients in the 200 subjects, we would expect 62 of these subjects to be discharged within 5 days without organ injury, and 54 subjects to have prolonged organ failure and/or late death. These numbers are well within the ranges required for statistical validation of these different models.

We anticipate that our overall consent rate for this observational study with minimal risk will be 75% meaning that to achieve an accrual rate of 25 trauma subjects per year at each institution, we will have to have 34 subjects per year meeting entry criteria. We expect no difficulty in accruing these 200 subjects over a four year period at the participating sites. They are both Level 1 trauma centers that have excess capacity to complete the proposed studies.

In this protocol, the only study specific intervention will be the collection of blood. The risks of drawing blood from a vein include discomfort at the site of puncture; possible bruising and swelling around the puncture site; rarely an infection; and, uncommonly, faintness from the procedure. Invasion of privacy will be negated with the use of coding for all data and specimens collected.

There are no direct benefits to study subjects for participation. This research may benefit society in the future. This study may one day result in new tests or treatments, or may help to prevent or cure diseases. No conflict of interest exists for the PI or sub-investigator.

ELIGIBILITY:
Inclusion Criteria Trauma Patients:

* All adults (age ≥18)
* Blunt trauma patients with hemorrhagic shock, defined by either a systolic BP (SBP) <90 mm Hg or base deficit (BD) <-6 meq
* Ability to obtain Informed Consent within 96 hours of injury.
* Ability to obtain the first lab draw within 12 hours of presentation to the Emergency Department.

Exclusion Criteria Trauma Patients:

* Patients not expected to survive greater than 48 hours.
* Patients with severe head injury.
* Severe pre-existing organ dysfunction
* Those that we are unable to obtain the first blood sample within 12 hours of injury
* Subjects who have received oncolytics within 14 days
* Subjects who are HIV + and have a CD4 count of <200/mm3
* Subjects not expected to survive 28 days due to pre-existing, uncorrectable medical condition
* Total body surface burns >40%
* Prisoners
* Current, chronic steroid use

If it is uncertain what the patient's past medical history is at the time of enrollment, they can be enrolled in the study and subsequently removed if they fail to meet criteria. This will be done because there are many circumstances with this patient population due to the severity of the injuries, the vulnerable nature of the patient at this early time, and the challenge in reaching the patient's legal representatives that we are unaware of their past medical history. The purpose of these exclusions is to ensure an adequate allocation of resources. Specifically, our goal is to evaluate patients at high risk for Multiple Organ Dysfunction Syndrome (MODS). Those with anticipated early death will add little to achieving this objective. Severe head injuries are excluded as well since the mortality in these subjects is usually attributable to their head injury rather than severe organ dysfunction. In addition, steroid use is known to affect the immunologic response to injury.

Inclusion Criteria Healthy Volunteers:

1. all adults (age ≥18)
2. Ability to obtain Informed Consent prior to blood collection.

Exclusion Criteria Healthy Volunteers:

1. Severe pre-existing organ dysfunction
2. Subjects who have received oncolytics within 14 days
3. Subjects who are HIV + and have a CD4 count of <200/mm3
4. Subjects not expected to survive 28 days due to pre-existing, uncorrectable medical condition
5. Total body surface burns >40%
6. Prisoners
7. Current, chronic steroid use

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2013-10; Primary Completion 2016-11 (Actual); Study Completion 2019-07-23 (Actual)

PRIMARY OUTCOMES:
Genomic score | Assement at the first 12 and 24 hours of hospitalization.
  A genomic score will be derived and assessed for each patient from the first two blood collections. A threshold score will be generated prior to the study initiation that will be used to statistically assign patients to either a "complicated outcome" or "other outcome", with primary goal being to identify severe trauma patients who are likely to have a complicated clinical course.
Time to recovery from organ injury. | Change in baseline through day 28 of the study.
  Time to recovery (TTR) is defined as the number of days in which the modified Marshall MODS score remains persistently above a score of zero. Designation of a "complicated outcome" is applied if the modified Marshall MODS score is above zero for greater than or equal to 14 days, or late death occurs. The designation of "other clinical outcome" will be a TTR less than 14 days.

SECONDARY OUTCOMES:
Mechanism of injury | Evaluated at the time of injury, information taken at baseline admission to emergency room.
  The circumstance in which an injury occurs, for example: sudden deceleration, wounding by a projectile, or crushing by a heavy object.
Initial hemodynamic variables | At baseline admission to emergency room.
  The first hemodynamic variables available following patient's admission to hospital.
Injury Severity Score | Obtained within 6 months following discharge from hospital.
  The Injury Severity Score (ISS) is an anatomical scoring system that provides an overall score for patients with multiple injuries. Each injury is assigned an Abbreviated Injury Scale (AIS) score and is allocated to one of six body regions (Head, Face, Chest, Abdomen, Extremities(including Pelvis), External). Only the highest AIS score in each body region is used. The 3 most severely injured body regions have their score squared and added together to produce the ISS score. The ISS score takes values from 0 to 75.
Patient demographics | Done at baseline admission to hospital.
  The patient's age, sex, race, ethnicity, height, weight, and BMI.
Time to definitive care | At baseline through the first 12 hours of admission to the hospital.
Total IV fluids received. | At baseline through the first 24 hours of admission to the hospital.
Type of IV fluids received | At baseline through the first 24 hours of admission to the hospital.
  Crystalloids and Colloids are considered IV fluids.
Plasma cytokines measured at time point number one | At baseline through the first 12 hours of admission to the hospital.
  Plasma cytokines will be measured by Luminex. The following cytokines will be determined: IL-6, IL-8, IL-10, IL-12p70, IL-15, IL-18, IL-23, GM-CSF, G-CSF, SDF-1, IP-10 (CXCL10), MCP-1, SDF-1 (CXCL12) and ckitL.
Plasma cytokines measured at time point number two. | Change in 12 hour to hour 24 after admission to the hospital.
  Plasma cytokines will be measured by Luminex™. The following cytokines will be determined: IL-6, IL-8, IL-10, IL-12p70, IL-15, IL-18, IL-23, GM-CSF, G-CSF, SDF-1, IP-10 (CXCL10), MCP-1, SDF-1 (CXCL12) and ckitL.
Overall incidence of ARDS | 48 hours after admission to the hospital through day 28 of the study.
  ARDS will be defined strictly based on the American-European Consensus Conference on ARDS published in 1994. Acute Lung Injury (ALI), a milder form of ARDS, will also be evaluated using the same clinical criteria except for a PaO2/FiO2 <300. The clinical research nurse will identify the development of ARDS and ALI by daily screening of the patients for these clinical criteria beginning 48 hours following injury.
Overall incidence of Multiple Organ Failure | 48 hours after admission to hospital through day 28 of the study.
  The development of additional organ dysfunction will be tracked by the well validated MOF Score (MOFScore). Its continuous nature allows detection of subtle differences in organ dysfunction not identified by dichotomous measures. The MOFscore assigns points to each of the six organ systems indicated and the summary score is calculated by summing the worst scores of each organ system over the course of the ICU stay. Because the MOFScore is designed to measure stable alterations in organ function, the first 48 hours post-injury are excluded. Those who die in first 48 hrs will be assigned the maximum MOF score of 24, and those who are discharged before 48 hrs will have a MOF score of 0.
  A score of 6 or greater will be considered MOF.
Mortality | Baseline through day 28 of the study.
  28 day mortality
Survival to hospital discharge. | Baseline admission to the hospital through discharge from the hospital.
Duration of hospital ICU stay | Baseline admission to the hospital through the last day in ICU.
Ventilator-free days | Baseline admission to the hospital through day 28 of the study.
Telephone Interview and Rand 36-Item Health Survey | Post hospital discharge at 4 months (+/- 60 days) and at 12 months (+/- 90 days)
  After discharge from the hospital for the trauma population, we will perform two post discharge telephone interviews to assess subject health and recovery. The first at 4 months (+/- 60 days) and the second at 12 months (+/- 90 days). The interviews will consist of a short questionnaire and the Rand 36-Item Health Survey 1.0.

OTHER OUTCOMES:
Nosocomial Infection | Baseline admission to the hospital through day 28 of the study.
  Central line-associated bloodstream infections, catheter-associated urinary tract infections, and ventilator-associated pneumonia. Infections may also occur at surgery sites, known as surgical site infections. Additionally, Clostridium difficile can cause gastrointestinal infection; patients can be exposed to this bacterium through contaminated surfaces or the spores can be transferred on unclean hands of others.
Resource Utilization and Mortality | Baseline admission to the hospital through day 28 in the study.

CONTACTS AND LOCATIONS:
Overall Officials: Lyle L Moldawer, Ph.D., Principal Investigator — University of Florida; Ronald Maier, M.D., Principal Investigator — University of Washington
Locations (2):
- United States (2):
  - UF Laboratory of Inflammation Biology and Surgical Science and Shands Hospital at UF, Gainesville, Florida
  - UW Harborview Research and Training Building, Seattle, Washington

REFERENCES:
- [Derived] Brakenridge SC, Wang Z, Cox M, Raymond S, Hawkins R, Darden D, Ghita G, Brumback B, Cuschieri J, Maier RV, Moore FA, Mohr AM, Efron PA, Moldawer LL. Distinct immunologic endotypes are associated with clinical trajectory after severe blunt trauma and hemorrhagic shock. J Trauma Acute Care Surg. 2021 Feb 1;90(2):257-267. doi: 10.1097/TA.0000000000003029. PMID 33214489
- [Derived] Mira JC, Cuschieri J, Ozrazgat-Baslanti T, Wang Z, Ghita GL, Loftus TJ, Stortz JA, Raymond SL, Lanz JD, Hennessy LV, Brumback B, Efron PA, Baker HV, Moore FA, Maier RV, Moldawer LL, Brakenridge SC. The Epidemiology of Chronic Critical Illness After Severe Traumatic Injury at Two Level-One Trauma Centers. Crit Care Med. 2017 Dec;45(12):1989-1996. doi: 10.1097/CCM.0000000000002697. PMID 28837430